CLINICAL TRIAL: NCT01787435
Title: A Cohort Study on the Association Between Acid-suppressing Drugs in Pregnancy and Asthma in the Offspring
Brief Title: Acid-suppressing Drugs Pregnancy Asthma Offspring Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9612N00018
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Asthma in Offspring
Keywords: Asthma,; acid-suppressing drugs,; pregnancy,; epidemiology
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- All women exposed to PPI at any time during pregnancy: Exposure to PPI defined as presence of at least one prescription of a PPI any time between last menstrual period and delievry date
  Interventions: Drug: Risk of asthma in offspring
- All women exposed to H2RA at any time during pregnancy: Exposure to H2RA defined as presence of at least one prescription of H2RA any time between last menstrual period and delivery date
  Interventions: Drug: Risk of asthma in offspring
- Pregnant women with no recorded use of acid suppressing drugs: Pregnant women with no recorded use of acid suppressing drugs at any time during pregnancy

INTERVENTIONS:
Drug: Risk of asthma in offspring — Exposure to PPI or H2RA, respectively during pregnancy
  No exposure to acid suppressing drugs during pregnancy
  Groups: All women exposed to H2RA at any time during pregnancy; All women exposed to PPI at any time during pregnancy

SUMMARY:
The purpose of this study is

1. To estimate the association between prenatal exposure to proton pump inhibitors (PPIs) and the risk of asthma during childhood.
2. To estimate the association between prenatal exposure to H2-receptor antagonists (H2RAs) and the risk of asthma during childhood.

DETAILED DESCRIPTION:
A cohort study on the association between acid-suppressing drugs in pregnancy and asthma in the offspring

ELIGIBILITY:
Inclusion Criteria:

- Females aged 18-45 years with at least one pregnancy between 1 January 1995 - 31 December 2010 (see study population description)

Exclusion Criteria:

- Males, females below age 18 and 45 years and above (see study population description)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women aged 18-45 years and with at least one pregnancy between 1 January 1995 and 31 December 2010 who have been enrolled with their PCP (Primary Care Physician) for at least 1 year and have had a health contact in the year prior to the last menstrual period (LMP) of the respective pregnancy. The final study population will include pregnancies that can be unequivocally linked with live birth(s) and only the first pregnancy ascertained during the study period for each woman will be retained
Sampling Method: Non-Probability Sample
Enrollment: 10116 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Relative risk of first asthma diagnosis associated with prenatal exposure to proton pump inhibitors | From 1 January 2005 till 31 December 2010, an expected average of 5 years.
Relative risk of first asthma diagnosis associated with prenatal exposure to histamine-2 receptor antagonists | From 1 January 2005 till 31 December 2010, an expected average of 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Garcia Rodriguez, MD, Principal Investigator — CEIFE (Centro Espanol de Investigacion Farmacoepidemiologica - Spanish Centre for Pharmacoepidemiologic Research )
Locations (1):
- Research Site, Madrid, Spain